CLINICAL TRIAL: NCT01684267
Title: Pelvic Obliquity Rehabilitation in Stroke Patients Using Robotically Generated Force Fields
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Northeastern University (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-000447
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Gait Re-training in Healthy Subjects; Gait Re-training in Stroke Survivors
Keywords: Stroke; Gait; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy (Experimental): Healthy individuals
  Interventions: Device: Robotic Gait Rehabilitation (RGR) Trainer
- Post-stroke (Experimental): Chronic stroke survivors
  Interventions: Device: Robotic Gait Rehabilitation (RGR) Trainer

INTERVENTIONS:
Device: Robotic Gait Rehabilitation (RGR) Trainer

SUMMARY:
To test the usability and effectiveness of a robotic device, called the Robotic Gait Rehabilitation (RGR) Trainer, in (1) healthy subjects with no gait impairment and (2) patients with stroke with gait abnormalities secondary to impaired knee function.

DETAILED DESCRIPTION:
The device is designed to train stroke patients to correct abnormal gait patterns associated with exaggerated and uncoordinated movements of the pelvis by applying force fields to correct the movement of the pelvis. The focus will be on correcting hip hiking (i.e. exaggerated unilateral upward movements of one side of the pelvis) in post-stroke patients. The human-robot interface will be based on impedance control techniques so that the force-field actuators generate smooth virtual spring/damper restitution forces at the patient's pelvic area.

As part of the study we will determine whether the force fields applied by the actuated components of the device can effect an acute change in gait biomechanics, primarily pelvis motion during stance and swing phases, in healthy subjects and patients with stroke during ambulation. The investigators will also evaluate the usability of the orthosis in terms of donning & doffing, user confidence, and comfort.

ELIGIBILITY:
HEALTHY

Inclusion Criteria:

* Can walk comfortably on a treadmill

Exclusion Criteria:

* any known orthopedic, musculoskeletal, neurological, cardiovascular, pulmonary, or gait disorder that results in an abnormal gait pattern
* Females in the second or third trimester of pregnancy

STROKE

Inclusion Criteria:

* single non-traumatic ischemic or hemorrhagic stroke at least 6 months prior to enrollment
* persistent hemiparesis, mild spasticity, and residual mild-to-moderate weakness of the lower extremity
* residual deficits of gait
* be able to ambulate without the use of assistive devices or assistance of a person
* able to walk at a comfortable walking speed of ~0.6 m/s
* able to walk safely on a treadmill
* medically stable
* No other neurological problems, or any known cardiovascular or musculoskeletal disorders that effects their gait or excludes them from exercise

Exclusion Criteria:

* unable to attend and follow instructions
* require physical assistance for ambulation
* other known orthopedic, musculoskeletal, neurological, cardiovascular, pulmonary, or gait disorder that results in an abnormal gait pattern
* severe joint contractures of the hemi-paretic knee
* females in the second or third trimester of pregnancy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pelvic obliquity | 1 day
  Change in pelvic obliquity during gait consequent to force application

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States